CLINICAL TRIAL: NCT02081391
Title: An Evaluation of the Efficacy and Safety of Tapentadol Oral Solution in the Treatment of Post-operative Acute Pain Requiring Opioid Treatment in Pediatric Subjects Aged From Birth to Less Than 18 Years Old
Brief Title: A Study to Look at Tapentadol Oral Solution in Children and Adolescents in Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Collaborators: Depomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KF5503/65; 2012-004359-35 (EudraCT Number)
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Acute Pain
Keywords: Acute Pain; Post-operative; Tapentadol; Opioid Treatment; Pediatric Participants
MeSH Terms: conditions — Acute Pain | interventions — Tapentadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial was double-blinded to prevent bias. The blind was broken for the participants aged 2 years to <18 years (Pediatric Committee of the European Medicines Agency [EU PDCO] set) before recruitment of the <6 month-old subjects for the United Sates Food and Drug Administration (US FDA) set (which comprised participants from birth to <18 years) was completed. Participants not belonging to the EU PDCO set (<2 years old) remained blinded (as independent randomization lists were used for participants aged <2 years old) and were unblinded only after the data base was locked for all participants from birth to <2 years old who were included in the US FDA <2 years population.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tapentadol immediate-release (IR) (Experimental): In the first 24 hours, tapentadol oral solution at a dose of 1.25 mg/kg body weight was given every 4 hours (±15 min) to participants aged 6 months to less than 18 years (maximum individual dose of tapentadol was 100 mg). Participants from 30 days to less than 6 months were dosed with 0.5 mg/kg body weight every 4 hours. Participants from birth to less than 30 days of age were dosed with 0.1 mg/kg body weight every 4 hours.
  After 24 hours and up to 72 hours, the dose could be reduced based on the investigator's judgment.
  Interventions: Drug: Tapentadol oral solution 4 mg/mL; Drug: Tapentadol oral solution 20 mg/mL
- Placebo (Placebo Comparator): Matching placebo oral solution was administered every 4 hours (±15 min) up to 72 hours.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tapentadol oral solution 4 mg/mL — Participants aged 6 months to less than 18 years old with a body weight below 20 kg received tapentadol oral solution 4 mg/mL by mouth every 4 hours for up to 72 hours.
  Participants from birth to less than 6 months received tapentadol oral solution, diluted 4 fold.
  Arms: Tapentadol immediate-release (IR)
Drug: Tapentadol oral solution 20 mg/mL — Participants aged from 6 months to less than 18 years with a body weight greater than or equal to 20 kg received tapentadol oral solution 20 mg/mL by mouth every 4 hours for up to 72 hours.
  Arms: Tapentadol immediate-release (IR)
Other: Placebo — Matching placebo oral solution was administered by mouth every 4 hours up to 72 hours.
  Arms: Placebo

SUMMARY:
The purpose of the study was to evaluate the efficacy of tapentadol oral solution, based on the total amount of supplemental opioid analgesic used over 12 hours or 24 hours after initiation of investigational medicinal product (IMP) in children and adolescents who had undergone surgery that would produce moderate to severe pain during opioid treatment.

DETAILED DESCRIPTION:
The supplemental opioid medication reflecting the standard of care was available as patient- or nurse-controlled intravenous (i.v.) morphine or hydromorphone. This supplemental opioid analgesic medication (SOAM) was given to control pain, as needed, in both the treatment and placebo groups.

Children and adolescents 6 months and older were dosed with a dose regimen of 1.25 mg/kg body weight for the first 24 hours of treatment. 24 hours after the start of study medication (and based on clinical judgment), a dose reduction to 1.0 mg/kg was allowed.

Participants 30 days to less than 6 months old were dosed with a regimen of 0.5 mg/kg for the first 24 hours of treatment. The dose of IMP could be reduced after 24 hours to 0.3 mg/kg (if there was a reduced need for analgesia according to the investigator's judgment).

Participants aged from birth to less than 30 days old were dosed with a regimen of 0.1 mg/kg for the first 24 hours of treatment. The dose of the IMP could be reduced after 24 hours to 0.075 mg/kg (if there was a reduced need for analgesia according to the investigator's judgment).

The decision to maintain or alter the dose based on the effectiveness of the analgesia (pain killer) and the adverse event profile observed in each participant over the first 24-hour dosing period was made based on the investigator's judgment.

In exceptional cases, if a participant had unbearable pain despite using nurse-controlled analgesia (NCA) or patient-controlled analgesia (PCA), an additional bolus (defined as a clinician bolus) of morphine or hydromorphone could have been administered. The clinician bolus could have been given either using the NCA/PCA pump system or by an intravenous bolus injection. The opioid given as a clinician bolus or if the NCA/PCA intravenous line failed, had to be the same opioid used in the NCA/PCA pump system.

Dosing with IMP was stopped if:

* A switch to exclusively oral opioid analgesic medication was indicated according to the local standard of care.
* Opioid analgesic medication was no longer needed.
* IMP had been administered for 72 hours.

Safety evaluations included assessment of adverse events, physical examination, vital signs, laboratory parameters, electrocardiogram, oxygen saturation, and, only for children older than 6 years of age, a scale to assess suicidal ideation (Columbia Suicide Severity Rating Scale [C-SSRS]). The maximum study duration for each participant was 42 days.

The evaluation of the safety and efficacy data was performed by age groups as aligned with European and United States agencies. Within the tapentadol treatment group, no analysis by tapentadol dose was conducted. Results for participants aged 2 years to <18 years were provided to the Pediatric Committee of the European Medicines Agency (EU PDCO) before recruitment of the children less than 6-month old required for the US Food and Drug Administration [FDA] analysis was completed. Participants from birth to <2 years old were analyzed separately for the US FDA only and not included in the analysis of the population aged from 2 years to <18 years.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent, and if applicable assent, given according to local regulations.
2. Male or female participant aged from birth (at least 37 weeks gestational age) to less than 18 years.
3. A female participant must be pre-menarchal, or surgically incapable of childbearing, or sexually abstinent, or if a female participant is sexually active, then she must be practicing an effective method of birth control (e.g., prescription hormonal contraceptives, intra-uterine devices used according to the product's instruction, double-barrier methods) before trial entry and throughout the trial.
4. A female participant must have a negative pregnancy test if aged 12 years or older, or is post-menarchal, or is sexually active.
5. Participant has undergone surgery (other than brain surgery or gastrointestinal surgery expected to affect the absorption of tapentadol [in the investigator's judgment]) that, in the investigator's opinion, would reliably produce moderate to severe pain requiring opioid treatment for at least 24 hours after first dose of IMP. Participants must remain hospitalized until the End of Treatment Visit.
6. Participant has received post-operative morphine or hydromorphone by NCA/PCA, with or without a background infusion of the same opioid, according to standard of care prior to allocation/randomization to IMP and participant is expected to require this morphine or hydromorphone by NCA/PCA after starting IMP.
7. Participant is able to tolerate liquids at the time of allocation/randomization to IMP.

Exclusion Criteria:

1. Participant, parent or the legal representative is an employee of the investigator or trial site, with direct involvement in the proposed trial or other trials under the direction of that investigator or trial site, or family member of the employees or the investigator.
2. Participant has been previously exposed to tapentadol.
3. Participant has received an experimental drug or used an experimental medical device within 28 days before allocation/randomization to IMP, or within a period less than 10 times the drug's half-life, whichever is longer.
4. Participant has a history or current condition of any one of the following:

   * Non-febrile seizure disorder.
   * Epilepsy.
   * Serotonin syndrome.
   * Traumatic or hypoxic brain injury, brain contusion, stroke, transient ischemic attack, intracranial hematoma, post-traumatic amnesia, brain neoplasm, or episode(s) of unconsciousness of more than 24 hours.
5. Participant has a history or current condition of any one of the following:

   * Moderate to severe renal or hepatic impairment.
   * Abnormal pulmonary function or clinically relevant respiratory disease (e.g., acute or severe bronchial asthma, hypercapnia).
6. Participant has a concomitant disease or disorder (e.g., endocrine, metabolic, neurological, psychiatric, infection, febrile seizure, paralytic ileus) that in the opinion of the investigator may affect or compromise participant safety during the study participation.
7. Participant has history of suicidal ideation or behavior.
8. Participant is obese in the investigator's judgment. Obesity can be determined based on appropriate body mass index (BMI) charts or tables; e.g., a BMI above the 97th percentile for children based on the World Health Organization growth charts or the participant's weight is less than 2500 grams.
9. Participant has a clinically relevant history of hypersensitivity, allergy, or contraindication to the supplemental opioid analgesic medication or tapentadol, or the excipients, or naloxone.
10. Participant is not able to understand and comply with the protocol as appropriate for the age of the participant or participant is cognitively impaired in the investigator's judgment such that they cannot comply with the protocol
11. Participant has a history of alcohol and/or substance abuse in the investigator's judgment based on participant's history and physical examination.
12. Participant is taking prohibited concomitant medication.
13. Participant has received a long-acting opioid for the treatment of pain following surgery within 6 hours of allocation/randomization to IMP.
14. Participant has clinically relevant (in the investigator's judgment) abnormal values for clinical chemistry or hematology (local laboratory sample taken after surgery).

    A participant aged 6 months to less than 18 years old is excluded if the:
    * Aspartate transaminase or alanine transaminase is greater 3-times upper limit of normal.
    * Total bilirubin is greater 2-times upper limit of normal (except if the cause is due to Gilbert's syndrome).
    * Glomerular filtration rate less than 60 mL/min.

    A participant aged from birth to less than 6 months old is excluded if:
    * Aspartate transaminase or alanine transaminase is >3-times upper limit of normal.
    * There is pathological jaundice in the opinion of the investigator.
    * Glomerular filtration rate (calculated according to Schwartz et al. 1984) is:

      * <20 mL/min/1.73 m2 for participants <1 week post-partum.
      * <30 mL/min/1.73 m2 for participants 1 week to 8 weeks post-partum.
      * <50 mL/min/1.73 m2 for participants >8 weeks postpartum to <6 months old.
15. Participant has:

    * Clinically relevant abnormal electrocardiogram (ECG).
    * Signs of pre-excitation syndrome.
    * Brugada's syndrome.
    * QT or corrected QT interval (QTc) interval >470 ms for children aged 6 years to less than 18 years old.
    * QT or QTc interval >460 ms for children aged from birth to less than 6 years old.
16. Peri- or post-operative analgesia supplied by a continuous regional technique (e.g., nerve block, wound infiltration catheter) or participant-controlled epidural analgesia that was terminated less than 6 hours before allocation/randomization to IMP.
17. Participant has post-operative clinically unstable systolic and diastolic blood pressure, heart rate, respiratory depression, or clinically unstable upper or lower airway conditions (in the investigator's judgment), or a saturation of peripheral oxygen (SpO2) <92% at the time of randomization (allocation/randomization to IMP).
18. Female participant is breast-feeding a child.
19. Participant requires continuous positive airway pressure or mechanical ventilation, at the time of allocation to IMP.
20. The mother of a newborn participant or the breastfeeding mother of a participant was administered a prohibited medication.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 216 (Actual)
Dates: Start 2015-02-19 (Actual); Primary Completion 2019-03-03 (Actual); Study Completion 2019-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (43):
- United States (13):
  - US008, Little Rock, Arkansas
  - US004, Stanford, California
  - US011, Miami, Florida
  - US012, Louisville, Kentucky
  - US001, The Bronx, New York
  - US018, The Bronx, New York
  - US006, Durham, North Carolina
  - US016, Cincinnati, Ohio
  - US015, Philadelphia, Pennsylvania
  - US014, Pittsburgh, Pennsylvania
  - US003, Dallas, Texas
  - US005, Houston, Texas
  - US007, Milwaukee, Wisconsin
- Bulgaria (3):
  - BG003, Pleven
  - BG005, Sofia
  - BG002, Stara Zagora
- Croatia (2):
  - HR003, Split
  - HR001, Zagreb
- Czechia (3):
  - CZ004, Fryštát
  - CZ003, Olomouc
  - CZ001, Praha 4 - Krč
- France (3):
  - FR002, La Tronche
  - FR001, Lille
  - FR004, Limoges
- DE001, Freiburg im Breisgau, Germany
- Hungary (2):
  - HU004, Budapest
  - HU003, Debrecen
- Poland (9):
  - PL011, Bydgoszcz
  - PL010, Gdansk
  - PL005, Lodz
  - PL002, Lublin
  - PL009, Olsztyn
  - PL014, Rzeszów
  - PL007, Torun
  - PL004, Warsaw
  - PL008, Warsaw
- Spain (5):
  - ES002, Barcelona
  - ES005, Madrid
  - ES007, Madrid
  - ES009, Santiago de Compostela
  - ES006, Valladolid
- United Kingdom (2):
  - GB003, Bristol
  - GB001, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Information available on the Grünenthal Web Site
Supporting Information: Study Protocol, SAP, CSR
URL: http://www.grunenthal.com/r-d-vision-mission/clinical-trials/data-sharing-clinical-trials

REFERENCES:
- [Background] Schwartz GJ, Feld LG, Langford DJ. A simple estimate of glomerular filtration rate in full-term infants during the first year of life. J Pediatr. 1984 Jun;104(6):849-54. doi: 10.1016/s0022-3476(84)80479-5. PMID 6726515

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial started on 19 Feb 2015 with the enrollment of the first participant. Recruitment of participants aged 2 to <18 years old was completed on 05 Dec 2016 with the last participant out. Recruitment of the remaining participants aged from birth to <2 years old was completed on 14 Mar 2019.
Pre-assignment Details: A total of 216 participants (or parents/caregivers) gave informed consent to participate in the trial, 180 of these participants were allocated to study drug (investigational medicinal product = IMP) and 175 participants received IMP (56 participants received placebo oral solution and 119 participants received tapentadol oral solution).
Groups:
- Tapentadol (From 2 to <18 Years): This arm includes all participants aged 2 years to less than 18 years who had undergone surgery that, in the investigator's opinion, would reliably produce moderate to severe pain requiring opioid treatment via NCA or PCA and who received at least 1 dose of tapentadol oral solution.
  12-hour treatment period completers were defined as participants who did not discontinue the treatment period before 12 hours. 24-hour treatment completers were defined as those who did not discontinue treatment before 24 hours; trial completers completed 24 hours of treatment and attended the follow up visit.
- Placebo (From 2 to <18 Years): This arm includes all participants aged 2 years to less than 18 years who had undergone surgery that, in the investigator's opinion, would reliably produce moderate to severe pain requiring opioid treatment via NCA or PCA and who received at least 1 dose of placebo oral solution.
  12-hour treatment period completers were defined as participants who did not discontinue the treatment period before 12 hours. 24-hour treatment completers were defined as those who did not discontinue treatment before 24 hours; trial completers completed 24 hours of treatment and attended the follow up visit.
- Tapentadol (From Birth to <2 Years): This arm includes all participants aged from birth (at least 37 weeks gestational age) to less than 2 years who had undergone surgery that, in the investigator's opinion, would reliably produce moderate to severe pain requiring opioid treatment via NCA and who received at least 1 dose of tapentadol oral solution.
  12-hour treatment period completers were defined as participants who did not discontinue the treatment period before 12 hours. 24-hour treatment completers were defined as those who did not discontinue treatment before 24 hours; trial completers completed 24 hours of treatment and attended the follow up visit.
- Placebo (From Birth to <2 Years): This arm includes all participants aged from birth (at least 37 weeks gestational age) to less than 2 years who had undergone surgery that, in the investigator's opinion, would reliably produce moderate to severe pain requiring opioid treatment via NCA and who received at least 1 dose of placebo oral solution.
  12-hour treatment period completers were defined as participants who did not discontinue the treatment period before 12 hours. 24-hour treatment completers were defined as those who did not discontinue treatment before 24 hours; trial completers completed 24 hours of treatment and attended the follow up visit.
Period: 12-hour Treatment
Arm/Group | Tapentadol (From 2 to <18 Years) | Placebo (From 2 to <18 Years) | Tapentadol (From Birth to <2 Years) | Placebo (From Birth to <2 Years)
Started | 108 | 52 | 11 | 4
Completed | 90 | 46 | 10 | 4
Not Completed | 18 | 6 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 0 | 0
Not completed — Physician Decision | 4 | 1 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 2 | 0 | 0
Not completed — Recovery (opioid no longer needed) | 2 | 0 | 1 | 0
Not completed — Further reasons | 2 | 1 | 0 | 0
Period: 24-hour Treatment and Trial Completion
Arm/Group | Tapentadol (From 2 to <18 Years) | Placebo (From 2 to <18 Years) | Tapentadol (From Birth to <2 Years) | Placebo (From Birth to <2 Years)
Started | 90 | 46 | 10 | 4
Completed | 63 | 28 | 9 | 4
Not Completed | 27 | 18 | 1 | 0
Not completed — Physician Decision | 10 | 5 | 0 | 0
Not completed — Lack of Efficacy | 1 | 3 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Recovery (opioid no longer needed) | 11 | 5 | 1 | 0
Not completed — Technical Problems | 1 | 1 | 0 | 0
Not completed — Further reasons | 3 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported separately for 160 participants aged 2 to less than 18 years (included in the Full Analysis Set for the EU PDCO and the US FDA) and for 15 participants aged from birth to less than 2 years (included in the Full Analysis Set for the US FDA). All participants completed 12 hours of treatment.
Groups:
- Tapentadol (From 2 to <18 Years) - 12-h Treatm. Completion: Participants had undergone surgery that, in the investigator's opinion, would reliably produce moderate to severe pain requiring opioid treatment via NCA or PCA.
  This arm includes all participants aged 2 years to less than 18 years who received at least 1 dose of tapentadol oral solution.
  12-hour treatment period completers were defined as participants who did not discontinue the treatment period before 12 hours.
- Placebo (From 2 to <18 Years) - 12-h Treatm. Completion: Participants had undergone surgery that, in the investigator's opinion, would reliably produce moderate to severe pain requiring opioid treatment via NCA or PCA.
  This arm includes all participants aged 2 years to less than 18 years who received at least 1 dose of placebo.
  12-hour treatment period completers were defined as participants who did not discontinue the treatment period before 12 hours.
- Tapentadol (From Birth to <2 Years) - 12-h Treatm. Completion: Participants had undergone surgery that, in the investigator's opinion, would reliably produce moderate to severe pain requiring opioid treatment via NCA.
  This arm includes all participants aged from birth (at least 37 weeks gestational age) to less than 2 years who received at least 1 dose of tapentadol oral solution.
  12-hour treatment period completers were defined as participants who did not discontinue the treatment period before 12 hours.
- Placebo (From Birth to <2 Years) - 12-h Treatm. Completion: Participants had undergone surgery that, in the investigator's opinion, would reliably produce moderate to severe pain requiring opioid treatment via NCA.
  This arm includes all participants aged from birth (at least 37 weeks gestational age) to less than 2 years who received at least 1 dose of placebo.
  12-hour treatment period completers were defined as participants who did not discontinue the treatment period before 12 hours.
- Total: Total of all reporting groups
Arm/Group | Tapentadol (From 2 to <18 Years) - 12-h Treatm. Completion | Placebo (From 2 to <18 Years) - 12-h Treatm. Completion | Tapentadol (From Birth to <2 Years) - 12-h Treatm. Completion | Placebo (From Birth to <2 Years) - 12-h Treatm. Completion | Total
Number analyzed (Participants) | 108 | 52 | 11 | 4 | 175
Age, Continuous [Mean (Full Range); unit: years] | 10.8 [2 to 17] | 10.4 [2 to 17] | 0.74 [0.1 to 1.6] | 0.48 [0.0 to 1.3] | 9.81 [0.0 to 17.0]
Age, Customized [Count of Participants; unit: Participants]
  Children (2 to <12 years) | 55 | 27 | 0 | 0 | 82
  Adolescents (12 to <18 years) | 53 | 25 | 0 | 0 | 78
  Birth to less than 28 days | 0 | 0 | 2 | 1 | 3
  28 days to less than 2 years | 0 | 0 | 9 | 3 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 23 | 5 | 2 | 83
  Male | 55 | 29 | 6 | 2 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 9 | 0 | 0 | 30
  Not Hispanic or Latino | 80 | 38 | 10 | 3 | 131
  Unknown or Not Reported | 7 | 5 | 1 | 1 | 14
Region of Enrollment [Number; unit: participants]
  Hungary | 4 | 3 | 1 | 1 | 9
  United States | 45 | 26 | 1 | 0 | 72
  Czechia | 7 | 3 | 0 | 0 | 10
  Poland | 20 | 5 | 9 | 2 | 36
  United Kingdom | 1 | 0 | 0 | 0 | 1
  Bulgaria | 10 | 5 | 0 | 0 | 15
  France | 3 | 3 | 0 | 0 | 6
  Germany | 4 | 2 | 0 | 0 | 6
  Croatia | 8 | 2 | 0 | 1 | 11
  Spain | 6 | 3 | 0 | 0 | 9
Height [Mean (Full Range); unit: centimeter] | 145 [87 to 185] | 143.3 [72 to 193] | 71.8 [54 to 84] | 65.3 [55 to 79] | 138.1 [54 to 193]
Weight [Mean (Full Range); unit: kg] | 43.09 [11.0 to 98.2] | 42.22 [10.7 to 89.1] | 7.97 [3.7 to 11.8] | 6.63 [3.9 to 11.3] | 39.79 [3.7 to 98.2]
Body Mass Index [Mean (Full Range); unit: kg per square meter] | 18.83 [9.5 to 29.7] | 19.12 [13.9 to 31.4] | 14.95 [11.0 to 17.8] | 14.73 [12.9 to 18.1] | 18.58 [9.5 to 31.4]
Amount of morphine or hydromorphone taken prior to IMP [Mean (Full Range); unit: mg/kg] | 0.59 [0.0 to 8.8] | 0.45 [0.0 to 3.7] | 0.26 [0.0 to 0.8] | 0.3 [0.2 to 0.4] | 0.52 [0.0 to 8.8]
Type of opioid analgesia used [Count of Participants; unit: Participants]
  Hydromorphone | 33 | 18 | 1 | 0 | 52
  Morphine | 75 | 34 | 10 | 4 | 123

OUTCOME MEASURES:

1. Primary Outcome: For the US FDA: The Total Amount of Supplemental Opioid Analgesic Medication Used Within the First 12 Hours After First Intake of Investigational Medicinal Product (IMP) [Tapentadol Oral Solution or Placebo]
Description: The primary endpoint for the United States Food and Drug Administration (US FDA) (and secondary endpoint for the Pediatric Committee of the European Medicines Agency [EU PDCO]) was the total amount of supplemental opioid analgesic medication (SOAM) used in the Full Analysis Set (from 2 years to <18 years old) within 12 hours after first intake of IMP. SOAM use is expressed in mg/kg of morphine i.v. equivalents.
Time Frame: Up to 12 hours
Population: Full Analysis Set; subset of 160 participants from 2 to less than 18 years included in the analysis. If by error a participant did not receive the allocated medication, the participant was evaluated as allocated following the intention-to-treat principle.
Measure: Least Squares Mean (Standard Error); unit: mg/kg
Groups:
- Tapentadol (From 2 to <18 Years): This analysis subset included all participants aged 2 years to less than 18 years old who were allocated to tapentadol and received at least one dose of IMP.
- Placebo (From 2 to <18 Years): This analysis subset included all participants aged 2 years to less than 18 years old who were allocated to placebo and received at least one dose of IMP.
Arm/Group | Tapentadol (From 2 to <18 Years) | Placebo (From 2 to <18 Years)
Number analyzed (Participants) | 108 | 52
mg/kg | 0.08 (0.01) | 0.13 (0.02)
Statistical Analysis 1: Comparison: Tapentadol (From 2 to <18 Years) vs Placebo (From 2 to <18 Years); The endpoint was analyzed using an analysis of variance model. This included treatment, baseline age group, and the used SOAM as factors. For participants discontinuing treatment before 12 hours for any other reason than no further need of opioid analgesics or switch to exclusively oral opioid analgesics, cumulative SOAM use over the respective time period was based on the observed SOAM use up to the time of the participant's discontinuation; Test type: Superiority; p = 0.0404, ANOVA; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.09 to 0], Standard Error of Mean 0.02

2. Primary Outcome: For the EU PDCO: The Total Amount of Supplemental Opioid Analgesic Medication Used Within the First 24 Hours After First Intake of IMP [Tapentadol Oral Solution or Placebo]
Description: The primary endpoint for the EU PDCO (and secondary endpoint for the US FDA) was the total amount of supplemental opioid analgesic medication (SOAM) used in the Full Analysis Set (from 2 years to <18 years old) within 24 hours after first intake of IMP. SOAM use is expressed in mg/kg of morphine i.v. equivalents.
Time Frame: Up to 24 hours
Population: Full Analysis Set; subset of 160 participants from 2 to less than 18 years included in the analysis; if by error a participant did not receive the allocated medication, the participant was evaluated as allocated following the intention-to-treat principle.
Measure: Least Squares Mean (Standard Error); unit: mg/kg
Arm/Group | Tapentadol (From 2 to <18 Years) | Placebo (From 2 to <18 Years)
Number analyzed (Participants) | 108 | 52
mg/kg | 0.14 (0.03) | 0.24 (0.03)
Statistical Analysis 1: Comparison: Tapentadol (From 2 to <18 Years) vs Placebo (From 2 to <18 Years); The endpoint was analyzed using an analysis of variance model. This included treatment, baseline age group, and the used supplemental opioid analgesic medication (SOAM) as factors. For participants discontinuing treatment before 24 hours for any other reason than no further need of SOAM or switch to exclusively oral opioid analgesics, cumulative SOAM use over the respective time period was based on the observed SOAM use up to the time of the participant's discontinuation; Test type: Superiority; p = 0.0154, ANOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.18 to -0.02], Standard Error of Mean 0.04

3. Secondary Outcome: Total Amount of Supplemental Opioid Analgesic Medication Received, Assessed in 12-hour Intervals From 24 Hours to 96 Hours After the First Dose of IMP
Description: The total amount of supplemental opioid analgesic medication (SOAM) received was assessed in 12-hour intervals from 24 hours to 96 hours after the first dose of IMP for participants who were administered SOAM.
  SOAM use was expressed in mg/kg of morphine i.v. equivalents.
Time Frame: Up to 96 hours
Population: Full Analysis Set; 175 participants aged from birth to <18 years; participants with no documented SOAM use in the respective time period are excluded from calculations. When 0 participants are indicated in the Row Analyzed that means no data was collected.
Measure: Mean (Full Range); unit: mg/kg
Groups:
- Tapentadol (From Birth to <2 Years): This analysis subset included all participants aged from birth to less than 2 years old who were allocated to tapentadol and received at least one dose of IMP.
- Placebo (From Birth to <2 Years): This analysis subset included all participants aged from birth to less than 2 years old who were allocated to placebo and received at least one dose of IMP.
Arm/Group | Tapentadol (From 2 to <18 Years) | Placebo (From 2 to <18 Years) | Tapentadol (From Birth to <2 Years) | Placebo (From Birth to <2 Years)
Number analyzed (Participants) | 108 | 52 | 11 | 4
mg/kg
  24 h to 36 h: number analyzed (Participants) | 38 | 19 | 1 | 1
  24 h to 36 h | 0.08 [0.0 to 0.4] | 0.14 [0.0 to 0.7] | 0.020 [0.02 to 0.02] | 0.003 [0.003 to 0.003]
  36 h to 48 h: number analyzed (Participants) | 30 | 12 | 1 | 1
  36 h to 48 h | 0.06 [0.0 to 0.4] | 0.06 [0.0 to 0.4] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]
  48 h to 60 h: number analyzed (Participants) | 20 | 8 | 0 | 0
  48 h to 60 h | 0.05 [0.0 to 0.4] | 0.06 [0.0 to 0.4] |  |
  60 h to 72 h: number analyzed (Participants) | 10 | 6 | 0 | 0
  60 h to 72 h | 0.06 [0.0 to 0.2] | 0.03 [0.0 to 0.2] |  |
  72 h to 84 h: number analyzed (Participants) | 3 | 2 | 0 | 0
  72 h to 84 h | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] |  |
  84 h to 96 h: number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Palatability of IMP After First Dose Assessed Using Facial 5-point Hedonic Scale
Description: Palatability of IMP after the first dose was assessed in participants aged 2 years to less than 18 years using 5-point hedonic scales in combination with verbal rating. A question "How does the medication taste" was asked and the verbal rating was from really good, good, a bit good/a bit bad, bad, and really bad. The pictorial scale of facial expressions was co-related with verbal rating range where 5 = really good, 4 = good, 3 = a bit good/a bit bad, 2 = bad, and 1 = really bad. Higher scores represent good palatability. Responses were summarized. Missing values were not imputed.
  Palatability data was not collected for participants <2 years old.
Time Frame: Up to 96 hours
Population: Full Analysis Set; subset of 160 participants aged from 2 years to less than 18 years included in the analysis. If by error a participant did not receive the allocated medication, the participant was evaluated as allocated following the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Tapentadol (From 2 to <18 Years) | Placebo (From 2 to <18 Years)
Number analyzed (Participants) | 108 | 52
Participants
  Really bad | 13 | 2
  Bad | 28 | 2
  A bit bad / a bit good | 36 | 10
  Good | 24 | 24
  Really good | 6 | 11
  Missing | 1 | 3

5. Secondary Outcome: Acceptability of IMP After First Dose Assessed Using Facial 5-point Hedonic Scale
Description: Acceptability of IMP in participants aged 2 years to less than 18 years was assessed using 5-point hedonic scales in combination with verbal rating. A question "Swallowing the medication is..." was asked and the verbal rating was from really good, good, a bit good/a bit bad, bad, and really bad. The pictorial scale of facial expressions was co-related with verbal rating range, with 5 = really easy, 4 = easy, 3 = a bit easy/a bit difficult, 2 = difficult, and 1 = really difficult. Higher scores represent better acceptability.
  Responses were summarized. Missing values were not imputed. Acceptability data was not collected in participants <2 years old.
Time Frame: Up to 96 hours
Population: Full Analysis Set: subset of 160 participants aged from 2 years to <18 years included in the analysis. If by error a participant did not receive the allocated medication, the participant was evaluated as allocated following the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Tapentadol (From 2 to <18 Years) | Placebo (From 2 to <18 Years)
Number analyzed (Participants) | 108 | 52
Participants
  Really difficult | 1 | 0
  Difficult | 7 | 3
  A bit difficult/a bit easy | 17 | 7
  Easy | 46 | 20
  Really easy | 35 | 19
  Missing | 2 | 3

6. Secondary Outcome: Change From Baseline in the Face, Leg, Activity, Cry, and Consolability (FLACC) Total Score in Participants Aged Less Than 6 Years
Description: The FLACC scale was used for children from birth to less than 6 years, or in older children who were not able to report their pain using the other scales. This tool includes 5 categories of pain behaviors: facial expression (F), leg movement (L), activity (A), cry (C), and consolability (C). Each of the 5 categories is scored 0, 1 or 2. The total score between 0 and 10 is the sum of the 5 individual categories. Higher scores represent worse condition.
  The Pain intensity scores were obtained before and after first dose of IMP, and before each subsequent dose of IMP, whenever possible, up to end of treatment (96 hours).
  Changes from baseline values were summarized descriptively for each time point.
Time Frame: Up to 96 hours
Population: Full Analysis Set: subset of 51 participants aged from birth to <6 years included in the analysis; participants with missing data were excluded from calculations. No standard deviations were derived for less than 5 participants.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Tapentadol (From 2 to <6 Years): This analysis subset included all participants aged 2 years to less than 6 years old who were allocated to tapentadol and received at least one dose of IMP.
- Placebo (From 2 to <6 Years): This analysis subset included all participants aged 2 years to less than 6 years old who were allocated to placebo and received at least one dose of IMP.
Arm/Group | Tapentadol (From 2 to <6 Years) | Placebo (From 2 to <6 Years) | Tapentadol (From Birth to <2 Years) | Placebo (From Birth to <2 Years)
Number analyzed (Participants) | 23 | 13 | 11 | 4
score on a scale
  30-60 mins after 1st IMP: number analyzed (Participants) | 22 | 13 | 11 | 4
  30-60 mins after 1st IMP | 1.1 [-5.0 to 4.0] | 1.9 [0.0 to 6.0] | 1.4 [-4.0 to 6.0] | 2.8 [0.0 to 5.0]
  Before 2nd dose of IMP | 1.4 [-2.0 to 7.0] | 1.3 [0.0 to 6.0] | 0.7 [-5.0 to 6.0] | 1.0 [0.0 to 2.0]
  Before 3rd dose of IMP: number analyzed (Participants) | 23 | 13 | 10 | 4
  Before 3rd dose of IMP | 1.7 [-2.0 to 7.0] | 1.6 [-1.0 to 6.0] | 2.0 [0.0 to 6.0] | -1.3 [-6.0 to 2.0]
  Before 4th dose of IMP: number analyzed (Participants) | 21 | 12 | 10 | 4
  Before 4th dose of IMP | 1.4 [-2.0 to 5.0] | 1.3 [-1.0 to 6.0] | 1.3 [-5.0 to 5.0] | 0.0 [-5.0 to 3.0]
  Before 5th dose of IMP: number analyzed (Participants) | 20 | 11 | 10 | 4
  Before 5th dose of IMP | 1.8 [-1.0 to 5.0] | 1.9 [-1.0 to 6.0] | 1.4 [-2.0 to 6.0] | 2.0 [0.0 to 4.0]
  Before 6th dose of IMP: number analyzed (Participants) | 19 | 8 | 10 | 4
  Before 6th dose of IMP | 1.6 [-2.0 to 5.0] | 2.3 [0 to 6.0] | 2.0 [-1.0 to 6.0] | 2.5 [0.0 to 5.0]
  Before 7th dose of IMP: number analyzed (Participants) | 19 | 8 | 8 | 3
  Before 7th dose of IMP | 1.6 [-2.0 to 6.0] | 2.1 [0.0 to 6.0] | 1.9 [-1.0 to 6.0] | 2.0 [0.0 to 3.0]
  Before 8th dose of IMP: number analyzed (Participants) | 13 | 5 | 5 | 2
  Before 8th dose of IMP | 1.2 [-1.0 to 4.0] | 2.2 [-3.0 to 6.0] | 3.8 [1.0 to 6.0] | -0.5 [-5.0 to 4.0]
  At End of Treatment | 2.4 [-3.0 to 6.0] | 2.0 [-1.0 to 9.0] | 2.1 [-4.0 to 6.0] | 3.5 [0.0 to 7.0]

7. Secondary Outcome: Change From Baseline Pain Intensity Using the Faces Pain Scale-Revised (FPS-R) in Participants Aged 6 to Less Than 12 Years
Description: For children aged 6 years (if possible) to less than 12 years, pain intensity was assessed by the use of the Faces Pain Scale-Revised (FPS-R). The FPS-R is a validated self-reported 6-point scale (0, 2, 4, 6, 8, 10) with 0 representing no pain and 10 representing very much pain. Facial representations were used to indicate how much the pain hurts. Higher scores represent worse condition.
  Pain intensity scores were obtained before and after first dose of IMP, and before each subsequent dose of IMP, whenever possible.
  Changes from baseline pain values were summarized descriptively for each time point up to end of treatment (96 hours).
Time Frame: Up to 96 hours
Population: Full Analysis Set: subset of 46 participants aged from 6 to less than 12 years included in the analysis; participants with missing data are not included in the analysis. If by error a participant did not receive the allocated medication, the participant was evaluated as allocated following the intention-to-treat principle.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tapentadol (6 to <12 Years): This analysis subset included all participants aged 6 years to less than 12 years old who were allocated to tapentadol and received at least one dose of IMP.
- Placebo (6 to <12 Years): This analysis subset included all participants aged 6 years to less than 12 years old who were allocated to placebo and received at least one dose of IMP.
Arm/Group | Tapentadol (6 to <12 Years) | Placebo (6 to <12 Years)
Number analyzed (Participants) | 32 | 14
units on a scale
  30-60 mins after 1st IMP: number analyzed (Participants) | 30 | 14
  30-60 mins after 1st IMP | 1.0 (1.72) | 0.7 (1.86)
  Before 2nd dose of IMP: number analyzed (Participants) | 27 | 12
  Before 2nd dose of IMP | 1.0 (2.5) | 0.5 (2.84)
  Before 3rd dose of IMP: number analyzed (Participants) | 26 | 12
  Before 3rd dose of IMP | 1.0 (2.35) | -0.2 (2.17)
  Before 4th dose of IMP: number analyzed (Participants) | 24 | 12
  Before 4th dose of IMP | 1.3 (2.33) | -0.3 (3.7)
  Before 5th dose of IMP: number analyzed (Participants) | 24 | 11
  Before 5th dose of IMP | 0.8 (2.75) | 0 (2.19)
  Before 6th dose of IMP: number analyzed (Participants) | 23 | 10
  Before 6th dose of IMP | 0.5 (2.43) | 0.2 (2.2)
  Before 7th dose of IMP: number analyzed (Participants) | 21 | 9
  Before 7th dose of IMP | 2.0 (2.37) | 0.7 (2.24)
  Before 8th dose of IMP: number analyzed (Participants) | 14 | 9
  Before 8th dose of IMP | 1.3 (2.55) | 0.2 (2.73)
  At End of Treatment | 2.8 (2.93) | 3.4 (3.56)

8. Secondary Outcome: Change From Baseline in the Visual Analog Scale (VAS) Pain Intensity Score in Participants Aged 12 to Less Than 18 Years
Description: For children and adolescents aged 12 years to less than 18 years, pain intensity was assessed by the use of a Visual analog scale (VAS). The participant was asked to draw a single line to indicate the current level of pain intensity on a 100 mm long scale by marking a point on the line in response to: "My pain right now is". The mark was scored between "no pain" and "pain as bad as it could be". A value of 0 indicates "no pain". A value of 100 indicates "pain as bad as it could be". Pain intensity scores were obtained before and after first dose of IMP, and before each subsequent dose of IMP, whenever possible. Changes from baseline values were summarized descriptively for each time point.
Time Frame: Up to 96 hours
Population: Full Analysis Set: subset of 78 participants aged from 12 to less than 18 years included in the analysis; participants with missing data are not included in the analysis. If by error a participant did not receive the allocated medication, the participant was evaluated as allocated following the intention-to-treat principle.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tapentadol (12 to <18 Years): This analysis subset included all participants aged 12 years to less than 18 years old who were allocated to Tapentadol and received at least one dose of IMP.
- Placebo (12 to <18 Years): This analysis subset included all participants aged 12 years to less than 18 years old who were allocated to placebo and received at least one dose of IMP.
Arm/Group | Tapentadol (12 to <18 Years) | Placebo (12 to <18 Years)
Number analyzed (Participants) | 53 | 25
units on a scale
  30-60 mins after 1st IMP: number analyzed (Participants) | 50 | 25
  30-60 mins after 1st IMP | 8.0 (18.67) | 6.4 (19.58)
  Before 2nd dose of IMP: number analyzed (Participants) | 48 | 24
  Before 2nd dose of IMP | 6.5 (23.61) | 6.0 (19.36)
  Before 3rd dose of IMP: number analyzed (Participants) | 44 | 22
  Before 3rd dose of IMP | 13.1 (25.09) | 5.9 (22.11)
  Before 4th dose of IMP: number analyzed (Participants) | 44 | 22
  Before 4th dose of IMP | 8.8 (29.01) | 5.1 (21.7)
  Before 5th dose of IMP: number analyzed (Participants) | 42 | 20
  Before 5th dose of IMP | 13.0 (22.92) | -2.7 (34.4)
  Before 6th dose of IMP: number analyzed (Participants) | 38 | 17
  Before 6th dose of IMP | 13.0 (24.74) | 6.6 (28.4)
  Before 7th dose of IMP: number analyzed (Participants) | 28 | 13
  Before 7th dose of IMP | 10.7 (25.77) | 15.0 (20.27)
  Before 8th dose of IMP: number analyzed (Participants) | 19 | 7
  Before 8th dose of IMP | 12.2 (28.91) | 11.9 (14.6)
  At End of Treatment: number analyzed (Participants) | 51 | 25
  At End of Treatment | 11.0 (27.87) | 11.4 (28.47)

9. Secondary Outcome: Clinical Global Impression of Change (CGIC)
Description: The CGIC was assessed at the End of Treatment Visit (Day 4). The investigator rated the participant's global improvement and satisfaction with the treatment on a 7-point scale with 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. Higher scores indicate worsening. Results were summarized descriptively.
Time Frame: Day 4
Population: Full Analysis Set; 175 participants from birth to less than 18 years are included. If by error a participant did not receive the allocated medication, the participant was evaluated as allocated following the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Tapentadol (From 2 to <18 Years) | Placebo (From 2 to <18 Years) | Tapentadol (From Birth to <2 Years) | Placebo (From Birth to <2 Years)
Number analyzed (Participants) | 108 | 52 | 11 | 4
Participants
  Very much improved | 15 | 12 | 3 | 1
  Much improved | 58 | 22 | 2 | 2
  Minimally improved | 18 | 8 | 1 | 1
  No change | 11 | 4 | 2 | 0
  Minimally worse | 3 | 2 | 1 | 0
  Much worse | 1 | 1 | 0 | 0
  Very much worse | 0 | 0 | 0 | 0
  Missing | 2 | 3 | 2 | 0

10. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: The PGIC was assessed at the End of Treatment Visit (Day 4). Participants rated their impression of overall status on a 7-point scale with 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. Higher scores indicate worsening. If participants were not capable of completing the questionnaire, the parent/legal guardian could completed the questionnaire on behalf of the participant.
  Results were summarized descriptively.
Time Frame: Day 4
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Tapentadol (From 2 to <18 Years) | Placebo (From 2 to <18 Years) | Tapentadol (From Birth to <2 Years) | Placebo (From Birth to <2 Years)
Number analyzed (Participants) | 108 | 52 | 11 | 4
Participants
  Very much improved | 16 | 11 | 4 | 3
  Much improved | 53 | 23 | 1 | 1
  Minimally improved | 21 | 12 | 1 | 0
  No change | 13 | 3 | 2 | 0
  Minimally worse | 1 | 0 | 0 | 0
  Much worse | 1 | 0 | 0 | 0
  Very much worse | 0 | 0 | 0 | 0
  Missing | 3 | 3 | 3 | 0

11. Secondary Outcome: Time to Receive First and Second Patient- or Nurse-controlled Analgesia After the First Dose of IMP
Description: The time to first and time to second patient-controlled analgesia (PCA) or nurse-controlled analgesia (NCA) after the first dose of IMP were summarized descriptively using time-to-event methods and are displayed by relevant treatment groups. Participants who completed the End of Treatment Visit (scheduled for 96 hours after first IMP) before their first/second use of NCA/PCA or participants who terminated treatment before their first/second use of NCA/PCA were censored at the End of Treatment Visit.
  Time-to-event variables are reported using Kaplan-Meier analyses. Therefore, values might remain missing if the survival function does not reach a respective threshold. This is indicated by not applicable (NA).
Time Frame: Up to 96 hours
Population: Full Analysis Set; 175 participants from birth to less than 18 years are included, censored participants are not displayed. If by error a participant did not receive the allocated medication, the participant was evaluated as allocated following the intention-to-treat principle.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Tapentadol (From 2 to <18 Years) | Placebo (From 2 to <18 Years) | Tapentadol (From Birth to <2 Years) | Placebo (From Birth to <2 Years)
Number analyzed (Participants) | 108 | 52 | 11 | 4
minutes
  Time to first NCA/PCA administration: number analyzed (Participants) | 81 | 46 | 6 | 3
  Time to first NCA/PCA administration | 183.0 [90.0 to 446.0] | 131.5 [74.0 to 216.0] | 960.0 [80.0 to NA] — Survival function did not reach threshold. | 155.0 [124.0 to NA] — Survival function did not reach threshold.
  Time to second NCA/PCA administration: number analyzed (Participants) | 66 | 37 | 4 | 1
  Time to second NCA/PCA administration | 572.0 [321.0 to 1993.0] | 388.0 [194.0 to 820.0] | NA [210 to NA] — Survival function did not reach threshold. | NA [500.0 to NA] — Survival function did not reach threshold.

12. Secondary Outcome: Time From First Dose of IMP Until Treatment Discontinuation Due to Lack of Efficacy
Description: The distributions of the time from the first dose of IMP to treatment discontinuation due to lack of efficacy were summarized descriptively using time-to-event methods.
  Participants who reached the maximum duration of treatment (72 hours) were censored at 72 hours after first IMP intake. Participants who discontinued during the Treatment Period for reasons other than lack of efficacy were censored at the time of the decision to discontinue treatment.
  Due to the low number of participants with events in the age group from 2 to <18 years, the median time and the corresponding confidence interval could not be calculated. The number of participants who discontinued early due to lack of efficacy is presented instead.
Time Frame: Up to 72 hours
Population: Full Analysis Set; 160 participants from 2 to less than 18 years were included in the analysis. If by error a participant did not receive the allocated medication, he/she was evaluated as allocated following the intention-to-treat principle. No participant <2 years was discontinued from treatment due to lack of efficacy; no analysis was performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Tapentadol (From 2 to <18 Years) | Placebo (From 2 to <18 Years) | Tapentadol (From Birth to <2 Years) | Placebo (From Birth to <2 Years)
Number analyzed (Participants) | 108 | 52 | 11 | 4
Participants
  Number of censored participants | 104 | 48 | 11 | 4
  Number of participants with event | 4 | 4 | 0 | 0

13. Secondary Outcome: Palatability of IMP After Last Dose Assessed Using Facial 5-point Hedonic Scale
Description: Palatability of IMP after the last dose in participants aged 2 years to less than 18 years was assessed using 5-point hedonic scales in combination with verbal rating. A question "How does the medication taste" was asked and the verbal rating was from really good, good, a bit good/a bit bad, bad, and really bad. The pictorial scale of facial expressions was co-related with verbal rating range with 5 = really good, 4 = good, 3 = a bit good/a bit bad, 2 = bad, and 1 = really bad. Higher scores represent good palatability. Responses were summarized. Missing values were not imputed.
  Palatability data was not collected in participants <2 years old.
Time Frame: Up to 96 hours
Population: Full Analysis Set; participants aged 2 to less than 18 years were included in the analysis. If by error a participant did not receive the allocated medication, the participant was evaluated as allocated following the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Tapentadol (From 2 to <18 Years) | Placebo (From 2 to <18 Years)
Number analyzed (Participants) | 108 | 52
Participants
  Really bad | 14 | 1
  Bad | 15 | 3
  A bit bad / a bit good | 38 | 14
  Good | 28 | 16
  Really good | 5 | 12
  Missing | 8 | 6

14. Secondary Outcome: Acceptability of IMP After Last Dose Assessed Using Facial 5-point Hedonic Scale
Description: as for outcome 5
Time Frame: Up to 96 hours
Population: Full Analysis Set; 160 participants aged 2 to less than 18 years were included in the analysis. If by error a participant did not receive the allocated medication, the participant was evaluated as allocated following the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Tapentadol (From 2 to <18 Years) | Placebo (From 2 to <18 Years)
Number analyzed (Participants) | 108 | 52
Participants
  Really difficult | 3 | 0
  Difficult | 6 | 2
  A bit difficult/a bit easy | 9 | 6
  Easy | 43 | 18
  Really easy | 39 | 20
  Missing | 8 | 6

15. Other Pre Specified Outcome: Mean Amount of Supplemental Opioid Analgesic Medication Use After First Intake of Investigational Medicinal Product in Children Aged From Birth to Less Than 2 Years
Description: The mean amount of supplemental opioid analgesic medication (SOAM) used in the Full Analysis Set subset aged from birth to less than 2 years old was determined from 0 to 12 hours and from 0 to 24 hours after first intake of IMP. SOAM use is expressed in mg/kg of morphine i.v. equivalents.
Time Frame: Up to 24 hours
Population: Full Analysis Set: subset of 15 participants from birth to less than 2 years included in the analysis; participants with missing data were excluded from calculations. If by error a participant did not receive the allocated medication, the participant was evaluated as allocated following the intention-to-treat principle.
Measure: Mean (Full Range); unit: mg/kg
Arm/Group | Tapentadol (From Birth to <2 Years) | Placebo (From Birth to <2 Years)
Number analyzed (Participants) | 11 | 4
mg/kg
  0-12 hours | 0.03 [0 to 0.07] | 0.01 [0 to 0.04]
  0-24 hours | 0.054 [0 to 0.3] | 0.016 [0 to 0.04]

16. Other Pre Specified Outcome: Median Amount of Supplemental Opioid Analgesic Medication Use After First Intake of Investigational Medicinal Product in Children Aged From Birth to Less Than 2 Years
Description: The median amount of supplemental opioid analgesic medication (SOAM) used in the Full Analysis Set subset aged from birth to less than 2 years old was determined from 0 to 12 hours and from 0 to 24 hours after first intake of IMP. SOAM use is expressed in mg/kg of morphine i.v. equivalents.
Time Frame: Up to 24 hours
Population: as for outcome 15
Measure: Median (Full Range); unit: mg/kg
Arm/Group | Tapentadol (From Birth to <2 Years) | Placebo (From Birth to <2 Years)
Number analyzed (Participants) | 11 | 4
mg/kg
  0-12 hours | 0.00 [0 to 0.07] | 0.01 [0 to 0.04]
  0-24 hours | 0.016 [0 to 0.3] | 0.013 [0 to 0.04]

ADVERSE EVENTS:
Time Frame: Any adverse event (AE) is reported that started at or after the first dose of IMP or started before the first dose of IMP and worsened in intensity after the first dose of IMP up to the end of the therapeutic reach of the last dose of IMP. The therapeutic reach is the time after IMP intake that a participant is still considered to be potentially affected by the study drug. For tapentadol oral solution, the therapeutic reach is defined as 48 hours.
Description: Adverse events are reported for all participants who received at least 1 dose of IMP (tapentadol or placebo) (Safety Set).
Groups:
- Overall (From 2 to <18 Years): All participants aged 2 years to below 18 years who received at least 1 dose of IMP.
- Tapentadol (From 2 to <18 Years): All participants aged 2 years to below 18 years who received at least 1 dose of tapentadol oral solution.
- Placebo (From 2 to <18 Years): All participants aged 2 years to below 18 years who received at least 1 dose of placebo oral solution.
- Overall (From Birth to <2 Years): All participants from birth to below 2 years who received at least 1 dose of IMP.
- Tapentadol (From Birth to <2 Years): All participants from birth to below 2 years who received at least 1 dose of tapentadol oral solution.
- Placebo (From Birth to <2 Years): All participants from birth to below 2 years who received at least 1 dose of placebo oral solution.
Arm/Group | Overall (From 2 to <18 Years) | Tapentadol (From 2 to <18 Years) | Placebo (From 2 to <18 Years) | Overall (From Birth to <2 Years) | Tapentadol (From Birth to <2 Years) | Placebo (From Birth to <2 Years)
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/108 | 0/52 | 0/15 | 0/11 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/160 | 2/108 | 0/52 | 0/15 | 0/11 | 0/4
Other Adverse Events (participants affected / at risk) | 87/160 | 61/108 | 26/52 | 9/15 | 6/11 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (From 2 to <18 Years) (N=160) | Tapentadol (From 2 to <18 Years) (N=108) | Placebo (From 2 to <18 Years) (N=52) | Overall (From Birth to <2 Years) (N=15) | Tapentadol (From Birth to <2 Years) (N=11) | Placebo (From Birth to <2 Years) (N=4)
Abdominal abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (From 2 to <18 Years) (N=160) | Tapentadol (From 2 to <18 Years) (N=108) | Placebo (From 2 to <18 Years) (N=52) | Overall (From Birth to <2 Years) (N=15) | Tapentadol (From Birth to <2 Years) (N=11) | Placebo (From Birth to <2 Years) (N=4)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site pruritus (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 11 (20) | 10 (19) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucinations, mixed (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Administration related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood urea decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 4 (5) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Po2 decreased (Investigations) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic anaemia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Painful Respiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 5 (8) | 4 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 6 (7) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 8 (8) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 17 (17) | 11 (11) | 6 (6) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 20 (27) | 16 (22) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 31 (44) | 25 (36) | 6 (8) | 2 (2) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lactic Acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
See primary endpoint for the US FDA.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves the right to review any proposed presentation of the results of this trial before they are submitted for publication or public disclosure. Neither party (e.g., the sponsor, the coordinating investigator) has the right to prohibit publication or public disclosure unless it can be shown to affect possible patent rights.

DOCUMENTS (2):
  • Study Protocol (2017-03-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT02081391/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT02081391/SAP_001.pdf